CLINICAL TRIAL: NCT05806580
Title: A Single-arm Prospective Study of Secondary Infusion of Relmacabtagene Autoleucel Injection for Relapsed or Refractory B-cell Lymphoma
Brief Title: Secondary Infusion of Relma-cel Injection for Relapsed or Refractory B-cell Lymphoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Vice president，Ruijin hospital, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JWCAR029019
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Relapsed or Refractory B-cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell | interventions — relmacabtagene autoleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relma-cel secondary infusion (Experimental)
  Interventions: Drug: Relma-cel

INTERVENTIONS:
Drug: Relma-cel — Patients who have undergone at least one disease assessment after initial Relma-cel treatment and have not achieved complete remission may receive a second treatment based on clinical practice. The specific dosage will be determined by the investigator according to the patient's condition and available dose reserves.
  Other Names: JWCAR029

SUMMARY:
To observe the efficacy and safety of a second infusion of relma-cel injection in patients with relapsed or refractory B-cell lymphoma.

DETAILED DESCRIPTION:
This study aims to collect efficacy and safety data from adult patients with relapsed or refractory large B-cell lymphoma (r/r LBCL) who receive a second infusion of relma-cel injection after initial treatment with relma-cel. The study will not include any form of grouping, and subgroup analysis will be conducted based on the actual data collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients have signed an Informed Consent Form (ICF).
* Adults diagnosed with relapsed or refractory B-cell lymphoma who have completed initial treatment with Relma-cel.
* Patients must have undergone at least one disease assessment post-initial Relma-cel treatment, and the investigator decides to administer a second treatment (including PR/PD/SD) based on clinical practice.
* Before the second infusion, confirm that the prepared dose of relma-cel is sufficient (recommended 80-150 x 10^6 CAR-T cells), with specific dosage determined by the investigator based on patient condition and dose availability.
* Confirm the presence of CD19+ residual tumor tissue, if clinically permissible.
* Measure plasma for the absence of anti-drug antibodies (ADA) to relma-cel before the second treatment.
* Toxicity related to lymphodepleting chemotherapy (fludarabine and cyclophosphamide), except for hair loss, must have resolved to ≤ Grade 1 or returned to baseline levels before retreatment.
* Patients must not have experienced severe adverse reactions during the first treatment, or any adverse reactions must have resolved to baseline levels from the first treatment.

Exclusion Criteria:

* Patients with hypersensitivity to active ingredients or any excipients (e.g., dimethyl sulfoxide, compound electrolyte injection, human albumin).
* Patients with uncontrolled systemic fungal, bacterial, viral, or other infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 3 months post CAR-T infusion
  ORR is defined as the percentage of participants achieving either CR or partial response (PR) per the Lugano Classification as determined by study investigators

CONTACTS AND LOCATIONS:
Locations (1):
- NO.197， Ruijin Er Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No